CLINICAL TRIAL: NCT04209842
Title: Utilization of Endoscopically Placed Intra-gastric Balloon in Obese and Morbid Obese Adolescents Combined With Behavioral Support
Brief Title: Effectiveness Gastric Balloon in Obese Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Roberto Gugig, professor of pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52936
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- gastric ballon placement (Experimental): will receive gastric balloon placed via endoscopy
  Interventions: Device: gastric balloon

INTERVENTIONS:
Device: gastric balloon — non surgical weight loss via placement of gastric balloon
  Other Names: Orbera

SUMMARY:
Assess the effectiveness of utilization of endoscopically placed intra-gastric balloon in obese and morbid obese adolescents combined with behavioral support for weight loss and health optimization.

ELIGIBILITY:
Inclusion Criteria:

* Clinically obese or morbid obese males and females aged 14 - 19 years old (BMI > 3.5 SD)
* Are able to attend biweekly to monthly sessions with our support team and are capable of adhering to the lifestyle changes advised

Exclusion Criteria

* Previous esophageal or gastric surgery or history of intestinal obstruction;
* History of moderate to severe inflammatory disease of the gastrointestinal tract such as esophagitis, gastric or duodenal ulcers or congenital anomalies such as atresias or stenosis; gastric or esophageal varices; congenital or acquired intestinal telangiectasis
* Hiatus hernia >5 cm or <5cm with associated severe or intractable gastro-esophageal reflux symptoms (assessed at balloon insertion);
* History of significant psychological disorder (permission sought from lead care giver).

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
change from baseline weight | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Gugig, MD, Principal Investigator — Stanford University; Monique T Barakat, MD, Principal Investigator — Stanford University
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No